CLINICAL TRIAL: NCT07238738
Title: Impact of Modified Periosteal Inhibition Technique on Alveolar Bone Stability in Immediate Implant Placement Procedures (Randomized Controlled Clinical Trial)
Brief Title: Comparison Between Modified Periosteal Inhibition (MPI) and Flapless Immediate Implant Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Meran Farid Hamza Awad, Assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPI with immediate implant
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Non-restorable Posterior Teeth; Thin Buccal Bone Plate; Buccal Bone Fenestraion
Keywords: Immediate Implant placement; Modified Periosteal Inhibition; Fenestration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flapless immediate implant placement with cortico-cancellous bone allograft in the gap distance (Experimental): Participants receive immediately inserted implant via flapless approach with the grafting of cortico-cancellous bone allograft in the gap distance between dental implant and surrounding native alveolar bone followed by insertion of customized healing abutment.
  Interventions: Procedure: Immediate implant placement via flapless approach
- Immediate implant placement with MPI technique using collagen sponge in gap distance (Experimental): Participants receive immediately inserted implant in conjunction with modified periosteal inhibition technique (MPI) after flap reflection from the buccal side and fixation of a 0.5 mm-thick cortical lamina glued to the buccal cortex with cyanoacrylate material. Collagen sponge will be filled in the gap distance followed by insertion of customized healing abutment.
  Interventions: Procedure: Immediate implant placement in conjunction with modified periosteal inhibition technique using collagen sponge in the gap distance
- Immediate implant with MPI technique using cortico-cancellous bone allograft in gap distance (Experimental): Participants receive immediately inserted implant in conjunction with MPI technique as described in group 2, however, cortico-cancellous bone allograft will be placed in the gap distance instead of collagen sponge and followed by insertion of customized healing abutment.
  Interventions: Procedure: Immediate implant placement in conjunction with modified periosteal inhibition technique using cortico-cancellous bone allograft in the gap distance

INTERVENTIONS:
Procedure: Immediate implant placement via flapless approach — Implant site preparation will be performed flapless using 3D computer assisted planned surgical stent. Implant site preparation will be performed using commercially available standard surgical kit. A single customized screw-type healing abutment will be screwed to the implant. Cortico-cancellous bone allograft will be inserted inside the extraction socket in the gap distance between the implant and surrounding alveolar bone of the fresh extraction socket.
  Arms: Flapless immediate implant placement with cortico-cancellous bone allograft in the gap distance
Procedure: Immediate implant placement in conjunction with modified periosteal inhibition technique using collagen sponge in the gap distance — After papillae incisions, an intra-sulcular incision will be made on the vestibular side of the extraction socket, extending to the mesial and distal mid-tooth with a #15c surgical scalpel. Implant site preparation will be performed using 3D computer assisted planned surgical stent. Implant site preparation will be performed using a standard surgical kit. A single customized screw-type healing abutment will be screwed to the implant. A full-thickness flap will be elevated creating a room that would allow the insertion of the cortical lamina. Cortical Lamina (0.5 mm thick) will be left in saline solution for 5 minutes and then cut to the desired shape, ranging from 8 to 10 mm in height, extending up to the mesial and distal margins of the extraction socket, molded until perfect fit and glued with two or three drops of N-butyl cyanoacrylate. A collagen sponge will be inserted inside the extraction socket to stabilize the clot. Suturing the papillae using 5-0 polypropylene monofilament.
  Arms: Immediate implant placement with MPI technique using collagen sponge in gap distance
Procedure: Immediate implant placement in conjunction with modified periosteal inhibition technique using cortico-cancellous bone allograft in the gap distance — After papillae incisions, an intra-sulcular incision will be made on the vestibular side of the extraction socket, extending to the mesial and distal mid-tooth with a #15c surgical scalpel. Implant site preparation will be performed using 3D computer assisted planned surgical stent. Implant site preparation will be performed using a standard surgical kit. A single customized screw-type healing abutment will be screwed to the implant. A full-thickness flap will be elevated creating a room that would allow the insertion of the cortical lamina. Cortical Lamina (0.5 mm thick) will be left in saline solution for 5 minutes and then cut to the desired shape, ranging from 8 to 10 mm in height, extending up to the mesial and distal margins of the extraction socket, molded until perfect fit and glued with two or three drops of N-butyl cyanoacrylate. cortico-cancellous bone allograft will be inserted in the gap distance. Suturing the papillae using 5-0 polypropylene monofilament.
  Arms: Immediate implant with MPI technique using cortico-cancellous bone allograft in gap distance

SUMMARY:
To clinically and radiographically assess the impact of the modified periosteal inhibition (MPI) technique, applied during immediate post-extraction implant placement, on alveolar bone dimensional changes, in comparison to the conventional flapless immediate implant approach.

DETAILED DESCRIPTION:
To assess the impact of the modified periosteal inhibition (MPI) technique, applied during immediate post-extraction implant placement in comparison to the conventional flapless immediate implant approach on radiographically by assessing marginal bone level measurements and bucco-lingual alveolar width. Clinically, pain levels, wound healing index, primary, secondary implant stability measured by resonance frequency analysis (RFA), peri-implant probing depth, and pink esthetic score (PES) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age ranges between 20 and 50 years including both genders.
* General good health (American Society of Anesthesiologists I-II).
* Presence of one hopeless non-restorable tooth requiring extraction at the posterior region.
* Adequate amount of palatal bone and basal bone (≥ 3 mm) to engage the immediately placed implants.
* Adequate keratinized soft tissue.
* Thick gingival phenotype (˃ 1.5 mm).
* Thin buccal bone plate or presence of fenestration.
* Favorable pattern of occlusion.
* Patient who is able to understand and sign a written consent.

Exclusion Criteria:

* Pregnancy or lactating females.
* Untreated periodontitis.
* Acute dentoalveolar infection.
* Complete absence of buccal bone plate.
* Osteometabolic disease.
* Chemotherapy or radiation therapy history of the neck-head area within the past 12 months.
* Heavy smokers (>20 cigarettes/per day) according to WHO.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation of horizontal and vertical dimensional changes of the alveolar bone placement by using cone beam computed tomography (CBCT). | Baseline, 6 months, 12 months after the implant placement
  1. Marginal Bone Level Measurements: It is the distance between a fixed reference point and the most apical point of connection between the implant surface and the bone. The reference point is the fixture-abutment interface.
  2. Bucco-lingual Alveolar Width: Width measurements will be made on tomographic slices perpendicular to the longitudinal axis of the alveolar crest at 1, 3 and 6 mm from summit of the alveolar crest.

SECONDARY OUTCOMES:
Pain Index | first post-operative day, third day and after one week.
  It will be evaluated using the Visual Analogue Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores represent worse outcomes.
Wound Healing Index (WHI) | 1 and 2 weeks after surgery
  score 1 indicates uneventful healing with no gingival edema, erythema suppuration, patient discomfort or flap dehiscence. Score 2 indicates uneventful healing with slight gingival edema, erythema, patient discomfort or flap dehiscence, but no suppuration. While score 3 indicates poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration.
Implant Stability Measurements | The RFA measurements will be made immediately after implant installation, and 3 months after implant placement before the prosthetic phase.
  The stability of the implant will be evaluated with resonance frequency analysis (RFA). The measurements will be made with the Osstell device by connecting the transducer (smart peg) to the fixture. The mesiodistal and buccolingual direction will be measured and the mean implant stability quotient will be determined.
Peri-implant Probing Depth (PPD) | Baseline, 6 months and 12 months post-operatively.
  Using a calibrated plastic periodontal probe, the distance between marginal border of the gingiva and the tip of the probe will be measured in mm.
Esthetic Evaluation | At the time of prosthetic phase (3 months after implant placement), 6 months, and 12 months postoperatively
  Esthetic scoring index called pink esthetic score (PES) index will be used in the current study. Seven variables will be scored; mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, alveolar process deficiency, soft tissue color, and texture of facial gingiva at the implant site. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. The mesial and distal papilla will be evaluated for completeness, incompleteness or absence. All other variables will be assessed by comparison with a reference tooth. The highest possible score reflecting a perfect match of the peri-implant soft tissue with that of the reference tooth will be 14. The PES index fulfilled important characteristics as inclusion of the peri-implant soft tissue and the restoration-inherent parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Meran F Awad, MSc, Principal Investigator — Mansoura University
Locations (1):
- Faculty of Dentistry, Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No